CLINICAL TRIAL: NCT04437745
Title: A Multicenter, Randomized, Rater-Blinded, No-Treatment Control Design Clinical Study to Evaluate the Effectiveness and Safety of YVOIRE Y-Solution 720 Injected Into the Mid-Face
Brief Title: To Evaluate the Effectiveness and Safety of YVOIRE Y-Solution 720 Injected Into the Mid-Face
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LG-HACL022
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Volume Defects in the Mid-face

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YVOIRE Y-Solution 720 (Experimental): Hyaluronic acid dermal filler
  Interventions: Device: YVOIRE Y-Solution 720
- Control (No Intervention): No Intervention

INTERVENTIONS:
Device: YVOIRE Y-Solution 720 — Hyaluronic acid dermal filler
  Arms: YVOIRE Y-Solution 720

SUMMARY:
To Evaluate the Effectiveness and Safety of YVOIRE Y-Solution 720 Injected Into the Mid-Face

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults 18 to 65 years of age (inclusive)
* 3 (moderate) or 4 (severe) on MFVDA-SRS
* sign the written informed consent form

Exclusion Criteria:

* have streptococcal disease or bleeding disorder
* have an active or infective skin disease, scars, or tumor on mid-face
* have congenital defect, trauma, abnormalities in adipose tissue related to immune-mediated diseases
* have undergone facial plastic surgery, tissue grafting, or tissue augmentation with silicone, fat, or other permanent, or semi-permanent procedures/treatment
* have undergone temporary facial dermal filler within 12 months, porcine-based collagen fillers within 24 months, or neuromodulator injections, mesotherapy, or resurfacing within 6 months
* have a medical history of hypertrophic cicatrix or keloid
* have radiation therapy experience on mid-face
* have a history of anaphylaxis, multiple severe allergies, atopy, or allergy to lidocaine, hyaluronic acid products, or Streptococcal protein

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Asian Faces Mid-Face Volume Deficit Severity Rating Scale (MFVDA-SRS) responder rate | 26 weeks from baseline
  the proportion of subjects with ≥1-grade reduction on the MFVDA-SRS score (The MFVDA-SRS score ranges from 1-4 with higher score indicating increasing severity of mid-face volume deficit.)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Wang, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China